CLINICAL TRIAL: NCT03018938
Title: Comparison Between Basal Insulin Analog and Insulin Analog Mid Mixture AS Starter Insulin for Chinese Patients With Type 2 Diabetes Mellitus (CLASSIC Study)
Brief Title: A Study of Basal Insulin Analog and Insulin Analog Mid Mixture in Chinese Participants With Type 2 Diabetes Mellitus
Acronym: CLASSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16507; F3Z-GH-IOQR (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-08-15

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: mid mixture insulin analog; basal insulin analog
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Analog Mid Mixture (Experimental): Insulin analog mid mixture given subcutaneously (SC).
  Interventions: Drug: Insulin Analog Mid Mixture
- Basal Insulin Analog (Experimental): Basal insulin analog given SC.
  Interventions: Drug: Basal Insulin Analog

INTERVENTIONS:
Drug: Insulin Analog Mid Mixture — Administered SC
  Arms: Insulin Analog Mid Mixture
Drug: Basal Insulin Analog — Administered SC
  Arms: Basal Insulin Analog

SUMMARY:
The purpose of this study is to compare the effectiveness of basal insulin analog and insulin analog mid mixture in Chinese participants with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* have type 2 diabetes as defined by World Health Organization (WHO) criteria
* are taking oral anti-hyperglycemic medications (OAMs) and are judged as OAM failure by the investigator
* most recent HbA1c value ≥7.5% within 12 weeks of study entry
* in the opinion of the investigator, require to initiate premix analog or basal insulin analog treatment
* willing to start with insulin treatment

Exclusion Criteria:

* have a diagnosis of type 1 diabetes
* have received any type of insulin within 24 months of study entry (except for intermittent use of insulin of less than 1 month each time)
* have serious preexisting medical or other conditions that, in the judgment of the investigator, would preclude participation in this study
* are pregnant or breastfeeding, or intend to become pregnant during the course of the study
* are currently enrolled or have participated, within the last 30 days in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- China (32):
  - Beijing Huaxin Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - China Meitan General Hospital, Chaoyang, Beijing Municipality
  - Beijing Yanhua hospital, Fangshan, Beijing Municipality
  - The 2nd Hospital of Lanzhou University, Lanzhou, Gansu
  - Shenzhen City People Hospital, Shenzhen, Guangdong
  - The 1st Hospital with Guangdong Pharmaceutical University, Yuexiu, Guangdong
  - The 1st Affiliated Hospital of Henan Science and technology, Luoyang, Henan
  - People's Hospital of Henan Province, Zhengzhou, Henan
  - Wuhan Union (Xiehe) Hospital, Wuhan, Hubei
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Nanjing TCM hospital, Nanjing, Jiangsu
  - Jiang Su Province Official Hospital, Nanjing, Jiangsu
  - Nanjing Jiangbei Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Taizhou City People Hospital, Taizhou, Jiangsu
  - The second People's hospital of Wuxi, Wuxi, Jiangsu
  - Xuzhou central Hospital, Xuzhou, Jiangsu
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Shanghai Pudong New Area Gongli Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New District Zhoupu Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Shunqing
  - The Third Affiliated Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Southwest Medical University Affiliated Hospital, Luzhou, Sichuan
  - Tianjin First Central Hospital, Nankai, Tianjin Municipality
  - Beijing LuHe Hospital Capital Medical University, Beijing, Tongzhou
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Peking University International Hospital, Beijing
  - Beijing Hai Dian Hospital, Beijing
  - Shanghai Yangpu District Central Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zeng T, Yuan H, Ren J, Li Y, Hou J, Du L, Zhu J, Chen L, Ji L. A Pragmatic Study of Basal and Mid-Mixture Insulins as Starter Insulins in Chinese Patients With Type 2 Diabetes: Observations From Long-Term, Real-World Experience. Diabetes Ther. 2021 Mar;12(3):931-941. doi: 10.1007/s13300-021-01007-z. Epub 2021 Feb 22. PMID 33616875

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Analog Mid Mixture: Participants received Insulin analog mid mixture given subcutaneously (SC) twice daily (BID) at the discretion of the investigator.
- Basal Insulin Analog: Participants received Basal insulin analog given subcutaneously (SC) once daily (QD) at the discretion of the investigator.
Period: Overall Study
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Started | 404 | 410
Received at Least 1 Dose of Study Drug | 404 | 410
Completed | 338 | 325
Not Completed | 66 | 85
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 21 | 32
Not completed — Withdrawal by Subject | 38 | 45
Not completed — Physician Decision | 3 | 2
Not completed — Sponsor Decision | 0 | 1
Not completed — Screen failure-After randomization | 4 | 2
Not completed — Not recorded | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Basal Insulin Analog: Participants received Basal insulin analog given subcutaneously (SC) once daily at the discretion of the investigator.
- Total: Total of all reporting groups
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog | Total
Number analyzed (Participants) | 404 | 410 | 814
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.8 (9.08) | 57.5 (9.29) | 57.6 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 177 | 358
  Male | 223 | 233 | 456
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 404 | 410 | 814
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 404 | 410 | 814
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 404 | 410 | 814
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 9.937 (1.6509) | 9.696 (1.5619) | 9.816 (1.6104)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by analysis of covariance (ANCOVA) model with last observation carried forward (LOCF) and with terms for change from baseline in HbA1c as response, treatment as fixed effect and baseline HbA1c as covariate.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for HbA1c.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 322 | 319
Percentage of HbA1c | -2.158 (0.0675) | -2.000 (0.0678)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Non-Inferiority — If Lower limit (L) >-0.4%, the Non-inferiority (NI) of basal insulin analog QD to insulin analog mid mixture BID is established; If Upper limit (U) <0.4%, the NI of insulin analog mid mixture BID to basal insulin analog QD is established; p = 0.1009, ANCOVA; LS Mean Difference (Final Values) = -0.158, 95% CI 2-sided [-0.346 to 0.031], Standard Error of Mean 0.0959

2. Secondary Outcome: Change From Baseline to Week 48 in HbA1c
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
  Least Squares (LS) mean was determined by ANCOVA model with LOCF and with terms for change from baseline in HbA1c as response, treatment as fixed effect and baseline HbA1c as covariate.
Time Frame: Baseline, 48 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 338 | 342
Percentage of HbA1c | -2.029 (0.0631) | -1.829 (0.0627)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0246, ANCOVA; LS Mean Difference (Final Values) = -0.201, 95% CI 2-sided [-0.376 to -0.026], Standard Error of Mean 0.0891

3. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <7% at Week 24
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: 24 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for HbA1c <7%.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 404 | 410
Percentage of participants | 33.9 | 28.3
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0941, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.95 to 1.87]

4. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <7% at Week 48
Description: as for outcome 3
Time Frame: 48 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 404 | 410
Percentage of participants | 23.3 | 23.4
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.8592, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.72 to 1.49]

5. Secondary Outcome: Change From Baseline to Week 24 in Venous Fasting Plasma Glucose
Description: Fasting Plasma glucose (FPG) is a test to determine how much glucose (sugar) is in a plasma sample after an overnight fast. Least Squares (LS) means was determined by ANCOVA model with LOCF and with terms for change from baseline in Venous FPG as response, treatment as fixed effect and baseline Venous FPG as covariate.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for Venous Fasting Plasma Glucose.
Measure: Least Squares Mean (Standard Error); unit: millimole/liter (mmol/L)
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 282 | 285
millimole/liter (mmol/L) | -2.332 (0.1525) | -2.755 (0.1517)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0497, ANCOVA; LS Mean Difference (Final Values) = 0.423, 95% CI 2-sided [0.000 to 0.846], Standard Error of Mean 0.2152

6. Secondary Outcome: Change From Baseline to Week 48 in Venous Fasting Plasma Glucose
Description: as for outcome 5
Time Frame: Baseline, 48 Weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: millimole/liter (mmol/L)
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 302 | 310
millimole/liter (mmol/L) | -2.527 (0.1391) | -3.174 (0.1373)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0010, ANCOVA; LS Mean Difference (Final Values) = 0.647, 95% CI 2-sided [0.263 to 1.031], Standard Error of Mean 0.1955

7. Secondary Outcome: Change From Baseline to Week 24 in Finger Stick Blood Glucose (FSBG)-Based Fasting Blood Glucose, Post Prandial Glucose
Description: Fasting blood glucose (FBG) and post prandial glucose (PPG) [pre-breakfast (fasting) and post-breakfast (approximately 2 hours after breakfast)] was measured using FSBG. LS Mean was measured with ANCOVA model with LOCF and with terms for change from baseline in FSBG-based FBG/PPG as response, treatment as fixed effect and baseline FSBG-based FBG/PPG as covariate.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for FBG and PPG.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 212 | 210
mmol/L
  FBG | -2.105 (0.1544) | -2.374 (0.1551)
  PPG: number analyzed (Participants) | 206 | 202
  PPG | -4.184 (0.2344) | -4.101 (0.2367)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; FBG; Test type: Superiority; p = 0.2193, ANCOVA; LS Mean Difference (Final Values) = 0.270, 95% CI 2-sided [-0.161 to 0.700], Standard Error of Mean 0.2191
Statistical Analysis 2: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; PPG; Test type: Superiority; p = 0.8014, ANCOVA; LS Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-0.739 to 0.571], Standard Error of Mean 0.3331

8. Secondary Outcome: Change From Baseline to Week 48 in Finger Stick Blood Glucose (FSBG)-Based Fasting Blood Glucose, Post Prandial Glucose
Description: as for outcome 7
Time Frame: Baseline, 48 Weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 237 | 232
mmol/L
  FBG | -2.233 (0.1429) | -2.724 (0.1444)
  PPG: number analyzed (Participants) | 231 | 226
  PPG | -4.372 (0.2129) | -4.359 (0.2153)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; FBG; Test type: Superiority; p = 0.0160, ANCOVA; LS Mean Difference (Final Values) = 0.491, 95% CI 2-sided [0.092 to 0.891], Standard Error of Mean 0.2033
Statistical Analysis 2: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; PPG; Test type: Superiority; p = 0.9661, ANCOVA; LS Mean Difference (Final Values) = -0.013, 95% CI 2-sided [-0.608 to 0.582], Standard Error of Mean 0.3028

9. Secondary Outcome: Total Daily Insulin Dose at Week 24 and 48
Description: Total daily insulin dose in the basal insulin analog and in Insulin Analog Mid Mixture group at week 24 and 48.
Time Frame: 24 Weeks, 48 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for Daily Insulin Dose.
Measure: Mean (Standard Deviation); unit: International Units (IU) per day
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 331 | 325
International Units (IU) per day
  24 Weeks | 24.89 (10.245) | 14.58 (7.093)
  48 Weeks: number analyzed (Participants) | 325 | 307
  48 Weeks | 24.22 (11.238) | 15.35 (7.090)

10. Secondary Outcome: Change From Baseline to Week 24 in Body Weight
Description: LS means were calculated using ANCOVA model with LOCF and with terms for change from baseline in bodyweight as response, treatment as fixed effect and baseline bodyweight as covariate.
Time Frame: Baseline, 24 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for Body Weight.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 356 | 366
kilograms (kg) | 1.226 (0.1976) | 0.559 (0.1949)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0166, ANCOVA; LS Mean Difference = 0.667, 95% CI 2-sided [0.122 to 1.211], Standard Error of Mean 0.2776

11. Secondary Outcome: Change From Baseline to Week 48 in Body Weight
Description: as for outcome 10
Time Frame: Baseline, 48 Weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 359 | 368
kilograms (kg) | 1.393 (0.2037) | 0.639 (0.2012)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.0086, ANCOVA; LS Mean Difference (Final Values) = 0.754, 95% CI 2-sided [0.192 to 1.316], Standard Error of Mean 0.2864

12. Secondary Outcome: Rate of Hypoglycemia at Week 24 and 48
Description: Hypoglycemic episodes are defined as events that are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 mmol/L). The overall yearly rates (events/participant/year) of those hypoglycemic events, calculated as, for each participant, the number of episodes times 365.25 and then divided by the participants treatment duration, will be summarized, and analyzed by a Negative-binomial regression model with treatment as fixed effects and log of (patient's treatment duration/365.25) as an offset variable.
Time Frame: 24 Weeks, 48 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for Hypoglycemia.
Measure: Mean (Standard Deviation); unit: Events/Participant/Year
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 124 | 76
Events/Participant/Year
  Nocturnal Hypoglycemia (24 Weeks): number analyzed (Participants) | 34 | 29
  Nocturnal Hypoglycemia (24 Weeks) | 0.54 (3.128) | 0.24 (0.955)
  Nocturnal Hypoglycemia (48 Weeks): number analyzed (Participants) | 42 | 38
  Nocturnal Hypoglycemia (48 Weeks) | 0.33 (1.931) | 0.20 (0.753)
  Total Hypoglycemia (24 Weeks): number analyzed (Participants) | 103 | 64
  Total Hypoglycemia (24 Weeks) | 1.60 (5.076) | 0.63 (1.785)
  Total Hypoglycemia (48 Weeks) | 1.18 (3.831) | 0.45 (1.188)

13. Secondary Outcome: Number of Participants With Insulin Treatment Change at Week 48
Description: Insulin treatment change can be insulin treatment discontinuation, switch, intensification or reduction in frequency.
  1. Discontinuation: Defined as stopping insulin treatment for 30 days or more.
  2. Switch: Defined as stop the initial insulin therapy and started another insulin therapy of different class.
  3. Intensification: Defined as any of the following: adding meal time insulin in basal insulin analog QD group; changing from BID to TID (Three times a day) in insulin analog mid mixture BID group
  4. Reduction in frequency: Defined as any of the following: changing from BID to QD; changing from TID to BID or QD.
Time Frame: Baseline through 48 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for Insulin Treatment Change.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 73 | 64
Participants
  Discontinuation | 23 | 31
  Switching | 23 | 24
  Intensification | 15 | 9
  Reduction | 12 | 0

14. Secondary Outcome: Percentage of Participants Who Achieve the HbA1c <7% Without Switching and Discontinuing Study Insulin, and Without Using Rescue Therapy at Week 24
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Percentages of participants who achieved HbA1c levels of <7% were analyzed using a logistic regression model with logic link function, treatment as fixed effect and baseline HbA1c as continuous covariate.
Time Frame: 24 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 404 | 410
Percentage of participants | 33.1 | 29.0
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.2009, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.89 to 1.77]

15. Secondary Outcome: Percentage of Participants Who Achieve the HbA1c <7% Without Switching and Discontinuing Study Insulin, and Without Using Rescue Therapy at Week 48
Description: as for outcome 14
Time Frame: 48 Weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 404 | 410
Percentage of participants | 23.9 | 23.7
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.8054, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.72 to 1.53]

16. Secondary Outcome: Change From Baseline to Week 48 in Self-Efficacy About Insulin Therapy Questionnaire (SEITQ) Score
Description: The SEITQ is designed to measure an individual's self-efficacy related to insulin therapy. The SEITQ consists of 5 items (that is, statements). The first 4 statements imply confidence in completing the tasks needed to take insulin correctly and avoid both hyperglycemia and hypoglycemia, whereas the last statement is an outcome expectation and implies that performance of these tasks will lead to avoidance of complications. Each item score ranges from 1 (strongly disagree) to 7 (strongly agree). The total SEITQ score is the sum of each item scores, with the range of 5 to 35. Higher SEITQ score indicates better outcome (higher self-efficacy). LS Mean was calculated using Mixed Models Analysis (MMRM) for repeated measures with all post-baseline SEITQ as responses, baseline SEITQ as a continuous covariate, treatment group, Visits, and treatment by visit interaction as fixed effects and participant as a random effect.
Time Frame: Baseline, 48 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline data for SEITQ Score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
Number analyzed (Participants) | 404 | 410
Units on a scale | -0.9 (0.23) | -0.8 (0.24)
Statistical Analysis 1: Comparison: Insulin Analog Mid Mixture vs Basal Insulin Analog; Test type: Superiority; p = 0.7553, Mixed Models Analysis; LS Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.5], Standard Error of Mean 0.33

ADVERSE EVENTS:
Time Frame: Up to 48 Weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | Insulin Analog Mid Mixture | Basal Insulin Analog
All-Cause Mortality (participants affected / at risk) | 0/404 | 1/410
Serious Adverse Events (participants affected / at risk) | 45/404 | 43/410
Other Adverse Events (participants affected / at risk) | 105/404 | 101/410
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Analog Mid Mixture (N=404) | Basal Insulin Analog (N=410)
Hyperglobulinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Rheumatic heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (3)
Diabetic retinopathy (Eye disorders) | 3 (3) | 2 (2)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (3) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 11 (11) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/223 (1) | 0/233 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Insulin Analog Mid Mixture (N=404) | Basal Insulin Analog (N=410)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Empty sella syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2)
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 8 (8) | 9 (9)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 4 (4) | 3 (3)
Diabetic retinopathy (Eye disorders) | 4 (4) | 5 (5)
Eyelid thickening (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Retinal vascular occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bowel movement irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysbiosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 3 (5) | 2 (2)
Swelling (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 4 (4)
Gallbladder polyp (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic calcification (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatic steatosis (Hepatobiliary disorders) | 11 (11) | 16 (16)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2)
Endometritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa fungal (Infections and infestations) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 2 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pulpitis dental (Infections and infestations) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinoscleroma (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Syphilis (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Trachoma (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 7 (7)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 3 (3)
Vaginal infection (Infections and infestations) | 3/181 (3) | 0/177 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/181 (0) | 1/177 (1)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Bone density decreased (Investigations) | 0 (0) | 1 (1)
Cardiothoracic ratio increased (Investigations) | 1 (1) | 0 (0)
Computerised tomogram liver abnormal (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 13 (13) | 9 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/181 (1) | 0/177 (0)
Carotid arteriosclerosis (Nervous system disorders) | 3 (3) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 9 (10) | 8 (8)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intellectual disability (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 5 (5) | 5 (5)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dyssomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 5 (5) | 3 (3)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 3 (4)
Nephropathy (Renal and urinary disorders) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal cyst (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/181 (1) | 0/177 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1/223 (1) | 0/233 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5/223 (5) | 8/233 (8)
Fallopian tube cyst (Reproductive system and breast disorders) | 0/181 (0) | 1/177 (1)
Menstruation irregular (Reproductive system and breast disorders) | 2/181 (2) | 0/177 (0)
Prostatic calcification (Reproductive system and breast disorders) | 1/223 (1) | 0/233 (0)
Prostatitis (Reproductive system and breast disorders) | 0/223 (0) | 2/233 (2)
Uterine cyst (Reproductive system and breast disorders) | 1/181 (1) | 0/177 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 4 (4) | 4 (4)
Diabetic vascular disorder (Vascular disorders) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 5 (5)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 3 (3)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 5 (5) | 4 (4)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-06-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03018938/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03018938/SAP_001.pdf